CLINICAL TRIAL: NCT06251674
Title: Comparison of Ultrasound-guided Transverse Carpal Ligament Needle Release Via Different Approaches for Patients With Mild-to-moderate Carpal Tunnel Syndrome
Brief Title: Efficacy of Ultrasound-guided Transverse Carpal Ligament Release for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhu Jiaan, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024PHB019-001
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: transverse carpal ligament; ultrasound; carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- long-axis group (Experimental): The patients in the long-axis group received one session of ultrasound-guided long-axis needle release of transverse carpal ligament.
  Interventions: Other: long-axis needle release
- short-axis group (Active Comparator): The patients in the short-axis group received one session of ultrasound-guided short-axis needle release of transverse carpal ligament.
  Interventions: Other: short-axis needle release

INTERVENTIONS:
Other: long-axis needle release — The participants received one session of ultrasound-guided long-axis TCL needle release.
  Arms: long-axis group
Other: short-axis needle release — The participants received one session of ultrasound-guided long-axis TCL needle release.
  Arms: short-axis group

SUMMARY:
Carpal tunnel syndrome (CTS) is one of the most common peripheral nerve entrapment neuropathies, and it is characterized by pain, numbness, tingling, and weakness in the regions innervated by the median nerve (MN). CTS is believed to result from compression of the MN as it passes through the narrowed carpal tunnel with regard to gradual ischemia and fibrosis.Ultrasound-guided needle release of transverse carpal ligament(TCL) is an effective method to decompress the carpal.There are two main approaches to perform the release, short-axis or long-axis. However, there is no consensus about the optimal strategy.Thus, this study aimed to compare the efficacy of these two approaches for patients with mild-to-moderate CTS.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* typical clinical signs of CTS present for at least three months, including pain, numbness, and tingling of the hands
* positive Phalen or Tinel sign
* electrophysiological parameters supportive of mild to moderate CTS
* high-resolution ultrasonography demonstrated MN compression at the carpal.

Exclusion Criteria:

* bifid MN or bilateral CTS
* pregnancy
* disorders such as rheumatic immune diseases, chronic renal failure, diabetes mellitus, hypothyroidism and other systemic diseases
* any accompanying disorder that could mimic CTS, such as thoracic outlet syndrome, cervical radiculopathy, polyneuropathy, proximal median nerve entrapment
* history of carpal tunnel surgery or injection into the affected carpal tunnel
* CTS caused by trauma, surgery, intracarpal lesions, or MN lesions malignant tumors or severe cardiorespiratory diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
visual analogue scale(VAS) scores | Baseline as well as 1 month, 3 month and 6 months after injection.
  The VAS scores is the most common tool to assess the level of pain. Possible scores range from 0(no pain) to 10(worst possible pain).

SECONDARY OUTCOMES:
Boston carpal tunnel syndrome questionnaire(BCTQ) | Baseline as well as 1 month, 3 month and 6 months after injection.
  BCTQ is the most commonly used evaluation for CTS symptoms; it contains two subscales: 11 items of symptom severity scale(SSS) and 8 items of functional status scale(FSS). Each item was scored 1-5 scores, with higher scores indicating greater severity and dysfunction.
cross-sectional area(CSA) of the median nerve | Baseline as well as 1 month, 3 month and 6 months after injection.
  CSA of the median nerve under ultrasound guidance reflects the severity of the disease to some extent

CONTACTS AND LOCATIONS:
Overall Officials: Jiaan Zhu, Dr, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wipperman J, Goerl K. Carpal Tunnel Syndrome: Diagnosis and Management. Am Fam Physician. 2016 Dec 15;94(12):993-999. PMID 28075090
- [Background] Orhurhu V, Orman S, Peck J, Urits I, Orhurhu MS, Jones MR, Manchikanti L, Kaye AD, Odonkor C, Hirji S, Cornett EM, Imani F, Varrassi G, Viswanath O. Carpal Tunnel Release Surgery- A Systematic Review of Open and Endoscopic Approaches. Anesth Pain Med. 2020 Dec 26;10(6):e112291. doi: 10.5812/aapm.112291. eCollection 2020 Dec. PMID 34150584
- [Background] Petrover D, Richette P. Treatment of carpal tunnel syndrome : from ultrasonography to ultrasound guided carpal tunnel release. Joint Bone Spine. 2018 Oct;85(5):545-552. doi: 10.1016/j.jbspin.2017.11.003. Epub 2017 Nov 16. PMID 29154980